# Inside Depression Clinical Trials: Patient Experiences Shared While Undergoing Clinical Trials

# Informed Consent Form (ICF) For <u>Power Clinical Trial's</u> Depression Observational Study

Date: June 30, 2023

Understanding the Informed Consent Document

Since you have been invited to consider participation in an observational clinical trial targeting individuals grappling with depression, you are given this informed consent form. It aims to provide a comprehensive account of the study's intricacies. This includes its overarching goals, the process, as well as a balanced portrayal of the potential advantages and disadvantages involved. Before making your decision, it is of utmost importance to thoughtfully deliberate your choices and seek guidance from a trusted confidant or your care team. In case any queries arise regarding the information presented, do not hesitate to approach the researcher for further clarification.

The Purpose Behind This Clinical Trial

Depression is a mental health disorder characterized by persistent feelings of sadness, loss of interest or pleasure in activities, and a range of other emotional and physical symptoms. It goes beyond normal fluctuations in mood and can significantly affect a person's daily functioning, relationships, and overall well-being.

The primary objective of conducting clinical trials for depression is to evaluate the safety and efficacy of emerging treatments. Through these trials, researchers strive to

determine the superiority of new treatments over existing ones, thereby gathering compelling evidence to endorse their utilization within the general populace.

This study seeks to delve into the firsthand experiences of patients diagnosed with depression who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

#### Significance of an Observational Clinical Trial

Embarking on this medical trial entails your involvement in an observational study—a distinctive type of clinical trial focused on gathering essential information by closely observing individuals, while upholding their existing care plans without any alterations.

Throughout the trial, researchers will diligently observe your journey and carefully measure the outcomes of your condition, abstaining from any intervention. Such trials serve as invaluable tools for acquiring a profound understanding of the inherent progression of a specific condition and its impact on individuals who receive a diagnosis. By actively participating in this observational study, you will make a meaningful contribution to the advancement of medical knowledge, thereby facilitating improvements in the care provided to individuals sharing the same condition.

# Comparing Depression Clinical Trials: An Exploration of Options

While the present clinical trial adopts an observational approach, refraining from administering specific treatments or interventions, it is crucial to acknowledge the existence of other clinical trials for depression that follow an interventional path, requiring participants to undergo targeted treatment regimens.

To make an informed decision about potential participation in a clinical trial, it is paramount to engage in comprehensive research and comparative analysis of different studies. Valuable information regarding <u>depression studies</u> can be obtained from clinicaltrials.gov or by visiting Power's website, which offers insights into ongoing <u>depression clinical trials</u> open for recruitment. By dedicating time and effort to understanding the various types of clinical trials available, you can confidently navigate your path and make a discerning choice regarding your suitability for trial participation.

#### Voluntary Participation in Surveys within a Clinical Trial

As a participant in this observational clinical trial, we value your input and aim to gather valuable insights into your experiences. This will be achieved through the completion of questionnaires every two weeks, requiring an estimated 20-30 minutes of your time. In addition, periodic check-in calls will be conducted on a quarterly basis for the duration of your participation in the trial.

It is essential to emphasize that your involvement in the survey component of this trial is entirely voluntary. You have the freedom to choose which questions to answer, and at any point, you may decide to discontinue your participation. We understand that the decision to participate in a clinical trial is personal, and we are committed to providing support throughout your journey. Your privacy and comfort are of utmost importance, and we will fully respect your decision-making process throughout the trial.

#### **Ensuring Anonymity in Survey Responses**

The confidentiality of your information is our utmost priority during this clinical trial. To ensure your anonymity, we kindly request that you refrain from including any personal or identifying details in your questionnaire responses. The research team will take all necessary precautions to protect your privacy. However, it is important to note that specific legal requirements may necessitate the disclosure of your data in certain circumstances.

# The Impact of Participation

Although immediate benefits may not be apparent for participants in this observational clinical trial, their involvement can have a profound impact on the lives of others. The data collected from participants will be instrumental in improving the enrollment process for future depression patients, streamlining their access to valuable medical research opportunities. By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future depression patients and play an active role in advancing medical research.

Safety and Risk Mitigation in Observational Trials

Clinical trials, while pivotal in medical advancements, may entail potential health risks, particularly when novel treatments are involved. However, it is important to note that our observational clinical trial eliminates such risks as participants are not subjected to any new interventions. Instead, participants are carefully observed, and outcomes are measured, ensuring their safety throughout the trial duration.

Preserving participant confidentiality is of utmost importance in clinical trials, and our medical study employs robust measures to ensure the privacy of participant information. All data collected from participants is anonymized, and access to this information is strictly restricted to the research team.

Moreover, comprehensive security protocols are implemented to safeguard all records, including call logs, online transactions, forms, and surveys. These records are securely stored using encryption and password protection, guaranteeing the confidentiality and protection of participant information. This stringent approach ensures that participant data remains confidential and shielded from unauthorized access, prioritizing the privacy and trust of all involved in the trial.

#### Participation Eligibility

We extend an invitation for your voluntary participation in an observational research study designed to explore the factors that drive patients' decisions to participate in clinical trials for depression. It is important to note that this study does not involve proposing new treatment protocols or making any changes to your current treatment plan.

Throughout this study, the researcher will conduct interviews to collect valuable information regarding your experiences. However, apart from the interviews, all aspects of your treatment and care will remain unchanged. The researcher will not provide a diagnosis or recommend any specific course of treatment. The primary objective of this study is to gather data for research purposes.

To be eligible for participation, it is necessary for you to be currently enrolled in another clinical trial for depression. By delving into the motivations behind your decision to participate and the factors influencing your determination to continue or discontinue treatment in that trial, we aim to gain deeper insights into patients' perspectives and experiences within clinical trials for depression.

Please remember that your participation in this study is entirely voluntary, and you have the freedom to withdraw at any time if you feel uncomfortable. Your decision to withdraw will not impact any of your legal rights, and your ongoing treatment plan in the other clinical trial will remain unaffected.

#### Further Exploration of Diversity in Clinical Trials

For those seeking a more in-depth understanding of representation in clinical trials, there is a plethora of online resources available to delve into this important topic. These resources offer valuable insights into the challenges and opportunities surrounding diversity in clinical research, providing a comprehensive perspective:

Masters, Joanna C., Jack A. Cook, Ginger Anderson, Gianluca Nucci, Anna Colzi, Marie-Pierre Hellio, and Brian Corrigan. "Ensuring diversity in clinical trials: The role of clinical pharmacology." *Contemporary Clinical Trials* 118 (2022): 106807.

Kahn, Justine M., Darrell M. Gray, Jill M. Oliveri, Chasity M. Washington, Cecilia R. DeGraffinreid, and Electra D. Paskett. "Strategies to improve diversity, equity, and inclusion in clinical trials." *Cancer* 128, no. 2 (2022): 216-221.

By engaging with these resources, individuals can gain valuable knowledge to inform their own involvement in clinical trials and actively contribute to promoting diversity and inclusivity in the field of medical research.

# Affirmation of Voluntary Participation

I affirm that I have dedicated ample time to thoroughly read and comprehend the informed consent form, either independently or with the assistance of a trusted individual who has read its contents to me. All of my inquiries and concerns have been adequately addressed to my complete satisfaction.

I am fully cognizant that my involvement in this study is entirely voluntary, and I possess the right to withdraw my consent at any time, without the need to provide a rationale or incur any financial obligations. I have been informed that a copy of this informed consent form will be provided to me for my personal records.

After careful contemplation and thoughtful consideration of all the information presented, I willingly consent to participate in this study of my own volition.

| Printed Name of Participant | |
|---|---|
| Participant Signature | |
| Date | |
| Confirmation by Consent Provider | |
| | th the contents of this document with the understanding of the purpose, methodologies, I aspects related to the depression clinical |
| and seek clarifications, effectively address have had. It is important to emphasize that | encourage the participant to ask questions sing any concerns or misconceptions they may at the participant's participation in this trial is nomy to withdraw their consent at any point, |
| Following their expression of consent, a consent for their personal reference. | opy of this document was furnished to the |
| Printed Name of Person Taking Consent | |
| Signature of Person Taking Consent | |
| Date | |